CLINICAL TRIAL: NCT02531191
Title: ASP015K Pharmacokinetic Study - Bioequivalence Evaluation of a Small and Current Tablet of ASP015K
Brief Title: Bioequivalence Evaluation of a New and Current Tablet of ASP015K
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 015K-CL-PK27
Record Dates: First submitted 2015-07-30; First posted 2015-08-24 (Estimated); Last update posted 2024-10-16 (Actual); Status verified 2019-09

CONDITIONS: Healthy Volunteers
Keywords: ASP015K; bioequivalence study; JAK inhibitor
MeSH Terms: interventions — peficitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- New Tablet Preceding Group (Experimental): Each subject received an ASP015K small tablet in period 1 and an ASP015K current tablet in period 2 under fasted conditions with 200 mL of water.
  Interventions: Drug: peficitinib
- Current Tablet Preceding Group (Experimental): Each subject received an ASP015K current tablet in period 1 and an ASP015K small tablet in period 2 under fasted conditions with 200 mL of water.
  Interventions: Drug: peficitinib

INTERVENTIONS:
Drug: peficitinib — oral
  Other Names: ASP015K

SUMMARY:
The objective of this study is to evaluate the bioequivalence of a new tablet versus a current tablet of ASP015K under fasting conditions after single oral administration in healthy male subjects.

DETAILED DESCRIPTION:
This is an open-label, randomized, single dose, 2-way crossover designed study. Forty non-elderly healthy male subjects will receive an ASP015K small tablet or an ASP015K current tablet in each period under fasted conditions. If the bioequivalence between two tablets cannot be demonstrated because of an insufficient number, an add-on subject study will be conducted as needed. The design of the add-on subject study will be the same with that of the initial study.

ELIGIBILITY:
Inclusion Criteria:

* 50.0 kg ≤ body weight at screening < 80.0 kg
* 17.6 ≤ BMI at screening < 26.4 [BMI = Body weight (kg) / (Body height (m))2]
* Subjects who agree to use the following highly effective contraception consisting of two forms of birth control (at least one of which must be a barrier method) starting at written informed consent through 90 days after the study drug administration in Period 2.
* Subjects who agree not to donate sperm starting at informed consent through 90 days after the study drug administration in Period 2.
* Subjects judged as healthy by investigator or sub-investigator based on physical examinations (subjective symptoms and objective findings) and all clinical tests obtained at screening and from check-in to immediately before the study drug administration in Period 1.

Exclusion Criteria:

* Subjects who have received investigational drugs within 120 days prior to screening or who plan to receive investigational drugs from screening assessment to check-in in Period 1 (Day -1).
* Any blood donation or blood drawing apply the following:

  * Whole blood collection (≥ 400 mL): from 90 days prior to screening to check-in in Period 1 (Day -1)
  * Whole blood collection (≥ 200 mL): from 30 days prior to screening to check-in in Period 1 (Day -1)
  * Platelet or plasma donation: from 30 days prior to screening to check-in in Period 1 (Day -1)
* Subjects who had used or plan to use any prescribed or non-prescribed drugs within 7 days prior to check-in in Period 1 (Day -1).
* Any deviation of blood pressure, pulse, body temperature, or 12-lead ECG at screening or check-in in Period 1 (Day -1) from the following normal range:

  * Supine pressure: Systolic: ≥ 90 mmHg, ≤ 140 mmHg; Diastolic: ≥ 40 mmHg, ≤ 90 mmHg
  * Supine pulse: ≥ 40 bpm, ≤ 99 bpm
  * Axillary temperature: ≥ 35.0 ºC, ≤ 37.0 ºC
  * 12-lead ECG: Normal or clinically irrelevant abnormality QTc interval: ≥ 330 msec, < 430 msec
* Any deviation of laboratory tests at Screening or on Day -1 (check-in) in Period 1 from the following normal range. Normal range of each test at the test or assay site will be used.

  * Hematology: > 20% of upper limit or < 20% of lower limit.
  * Chemistry: deviation of ALT, AST, Cre, blood electrolytes (Na, K, Cl), or fasting blood glucose. > 20% of upper limit or < 20% of lower limit in other than above tests; however no lower limit is set with respect to ALT, AST, γ-GTP, T-Bil, ALP, LDH, CK, T-Cho, TG, Cre, and UA.
  * Urinalysis (qualitative): deviation in any of the urinalysis.
  * Urinary drug abuse test: positive for benzodiazepines, cocaine-based narcotics, analeptic drugs, cannabis, barbituric acid derivatives, morphine-based narcotics, phencyclidines, or tricyclic antidepressants.
  * Immunological test: positive for HBs antigen, HBc antibody, HCV antibody, HIV antigen or antibody, or syphilis.
* Subjects who have any history or complication of drug allergies.
* Subjects who have a history of upper gastrointestinal symptoms, i.e. nausea, vomit, stomach ache, etc. within 7 days prior to check-in in Period 1 (Day -1).
* Subjects who have any history or complication of hepatic disease, i.e. viral hepatitis, drug induced liver injury, hepatic dysfunction, etc.
* Subjects who have any history or complication of cardiac disease, i.e. congestive heart failure, angina, arrhythmia requires a treatment, etc.
* Subjects who have any history or complication of respiratory disease, i.e. bronchial asthma, chronic bronchitis, pneumonitis, etc. (except for a history of asthma in childhood)
* Subjects who have any history or complication of gastrointestinal disease, i.e. peptic ulcer, reflux esophagitis, etc. (except for a history of appendicitis)
* Subjects who have any history of gastrointestinal resection (except for a history of appendectomy)
* Subjects who have any history or complication of renal disease, i.e. acute renal failure, glomerulonephritis, intestinal nephritis, etc.
* Subjects who have any history or complication of endocrine disease, i.e. hyperthyroidism, abnormality of growth hormone, etc.
* Subjects who have any history or complication of cerebrovascular disorder, i.e. cerebral infarction.
* Subjects who have any history or complication of malignant tumor.
* Subjects who have any history or complication of congenital short QT syndrome.
* Subjects who have any history or complication of lymphatic disease, i.e. lymphoproliferative disease.
* Subjects any of the following apply regarding tuberculosis:

  * History of active tuberculosis
  * Abnormality in chest X-ray test at screening
  * Contact with patients with infectious tuberculosis
* Subjects any of the following apply regarding infectious disease other than tuberculosis:

  * History or complication of serious herpes zoster or disseminated herpes zoster
  * More than once relapse of localized herpes zoster
  * Hospitalization due to serious infection within 90 days before check-in in Period 1 (Day -1)
  * I.V. antibiotics treatment within 90 days before check-in in Period 1 (Day -1) (except for prevention use)
  * Judged as prone to infections by investigator or sub-investigator, i.e. subjects with urethral catheterization.
* Subjects who have any history of inoculation of live vaccine or attenuated live vaccine within 56 days prior to check-in in Period 1 (Day -1).
* Subjects who have any history of clinically serious allergy (Clinically serious allergy; allergy induced systemic urticaria or anaphylactic shock require hospitalization when exposed to specific antigens or drugs).
* Subjects who have any history or complication of heart failure classified as NYHA Class III or IV.
* Subjects who have a history of ASP015K administration.
* Subjects with excessive alcohol drinking or smoking.

  * Criteria for "excessive":

    1. Smoking: ≥ 20 cigarettes/day
    2. Alcohol drinking: ≥ 45 g/day (a large bottle of beer contains 25 g of alcohol, 1 gou of Japanese sake contains 22 g of alcohol)
* Employee of the sponsor, CROs or study site involved in this study.
* Subjects judged as inappropriate for the study by investigator or sub-investigators.

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06-21 (Actual); Primary Completion 2015-07-15 (Actual); Study Completion 2015-07-15 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) parameter of ASP015K: Area under the concentration-time curve (AUC) from the time of dosing to the time of the last sampling (AUCt) | Up to 72 hours after each study drug dosing
Pharmacokinetics (PK) parameter of ASP015K: Maximum concentration (Cmax) | Up to 72 hours after each study drug dosing

SECONDARY OUTCOMES:
Safety assessed by Adverse Events (AEs) | Up to 6 days after the study drug dosing of Period 2
Safety assessed by Vital signs | Up to 6 days after the study drug dosing of Period 2
  Vital signs include systolic and diastolic blood pressures, pulse rate and temperature.
Safety assessed by Laboratory tests | Up to 6 days after the study drug dosing of Period 2
  Laboratory tests include hematology, biochemistry, urinalysis.
Safety assessed by 12-lead ECGs | Up to 6 days after the study drug dosing of Period 2
  12-lead ECG: 12-lead electrocardiogram
Pharmacokinetics (PK) profile of ASP015K: AUCinf | Up to 72 hours after each study drug dosing
  AUCinf: AUC from the time of dosing extrapolated to time infinity
Pharmacokinetics (PK) profile of ASP015K: AUClast | Up to 72 hours after each study drug dosing
  AUClast: AUC from the time of dosing to the last measurable concentration
Pharmacokinetics (PK) profile of ASP015K: CL/F | Up to 72 hours after each study drug dosing
  CL/F: Apparent total systemic clearance
Pharmacokinetics (PK) profile of ASP015K: kel | Up to 72 hours after each study drug dosing
  kel: Terminal elimination rate constant
Pharmacokinetics (PK) profile of ASP015K: MRTinf | Up to 72 hours after each study drug dosing
  MRTinf: Mean residence time from the time of dosing extrapolated to time infinity
Pharmacokinetics (PK) profile of ASP015K: t1/2 | Up to 72 hours after each study drug dosing
  t1/2: Terminal elimination half-life
Pharmacokinetics (PK) profile of ASP015K: tmax | Up to 72 hours after each study drug dosing
  tmax: Time of Cmax (Maximum concentration)
Pharmacokinetics (PK) profile of ASP015K: Vz/F | Up to 72 hours after each study drug dosing
  Apparent volume of distribution during the terminal elimination phase

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Toyoshima J, Shibata M, Kaibara A, Kaneko Y, Izutsu H, Nishimura T. Population pharmacokinetic analysis of peficitinib in patients with rheumatoid arthritis. Br J Clin Pharmacol. 2021 Apr;87(4):2014-2022. doi: 10.1111/bcp.14605. Epub 2020 Dec 1. PMID 33068028
- [Derived] Shibata M, Toyoshima J, Kaneko Y, Oda K, Kiyota T, Kambayashi A, Nishimura T. The Bioequivalence of Two Peficitinib Formulations, and the Effect of Food on the Pharmacokinetics of Peficitinib: Two-Way Crossover Studies of a Single Dose of 150 mg Peficitinib in Healthy Volunteers. Clin Pharmacol Drug Dev. 2021 Mar;10(3):283-290. doi: 10.1002/cpdd.843. Epub 2020 Jul 3. PMID 32618438